CLINICAL TRIAL: NCT05724797
Title: A Phase 1, First in Human, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study of NRS 033 in Healthy Volunteers
Brief Title: Single Ascending Dose Study of NRS 033 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nirsum Labs (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NRS-033-102; UG3DA048234 (NIH)
Record Dates: First submitted 2023-02-01; First posted 2023-02-13 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NRS-033: Cohorts 1-3 (Experimental): Cohorts 1-3: 6 participants in each cohort will receive active drug (NRS-033)
  Interventions: Drug: NRS-033
- Placebo: Cohorts 1-3 (Placebo Comparator): Cohorts 1-3: 2 participants in each cohort will receive the matching placebo dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NRS-033 — A single dose of NRS-033 will be administered
  Arms: NRS-033: Cohorts 1-3
Drug: Placebo — A single dose of matching placebo will be administered
  Arms: Placebo: Cohorts 1-3

SUMMARY:
This is a phase 1, first in human, randomized, double-blind, placebo-controlled, single ascending dose (SAD) study in healthy adult male and female subjects 18 to 55 years of age, inclusive.

DETAILED DESCRIPTION:
Subjects will provide written informed consent and undergo a screening visit within 28 days of receiving study drug. Eligible subjects must have a negative urine drug screen (UDS) and a negative naloxone challenge test at Screening and at the check-in visit (Day -1). Upon completion of screening, eligible subjects will be admitted to the clinical research unit (CRU) on Day -1 and remain confined in the CRU through completion of all scheduled procedures on Day 4 to allow for safety labs, pharmacokinetic (PK) blood draws, ECGs, injection site assessments, and adverse event monitoring.

Study medication dosing will occur in the morning on Day 1 and serial blood samples for plasma concentration determination for PK analysis will be taken during this time at pre-dose and 0.25, 0.50, 1, 1.5, 2, 4, 8, 10, 12, 24 (day 2), 48 (day 3), and 72 (day 4) hours post dose. Additional blood PK samples will be taken at follow-up visits. A Safety Review Committee (SRC) will review blinded, preliminary data from Cohort 1 to make recommendations regarding escalation to Cohorts 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 and ≤55 years of age at time of consent
* Body mass index ≥18.0 to ≤35.0 kg/m2
* Medically healthy based on the absence of clinically significant abnormal vital sign
* Females must have a negative serum pregnancy test at time of screening and negative urine pregnancy test upon admission; also, females of childbearing potential must agree to use a highly effective means of contraception from Screening until 9 months after receiving the study medication.
* Male subjects with female partners of childbearing potential must agree to use a male condom and will be advised of the benefit for a female partner to use a highly effective method of contraception
* Agree to stay within National Institute on Alcohol Abuse and Alcoholism (NIAAA) low risk drinking criteria. For women, low-risk drinking is no more than 3 drinks on any single day and no more than 7 drinks per week. For men, it is defined as no more than 4 drinks on any single day and no more than 14 drinks per week.
* Agree not to take opioid analgesics.

Exclusion Criteria:

* Clinically significant medical or psychiatric diagnosis (assessed on history, physical exam, ECG, and/or blood tests; includes significant history of cardiovascular, pulmonary, hepatic, gallbladder, or biliary tract, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychiatric disease, or active sexually transmitted disease).
* Significant neuropsychiatric diagnosis (e.g., major depression, suicidal ideation, multiple sclerosis, dementia) as reported by the subject, or a past history of suicide attempt.
* Females who are pregnant, lactating, or likely to become pregnant during the study.
* History over last 30 days of consuming alcohol >3 drinks day per day or >7 drinks per week if female; if male >4 drinks per day or >14 drinks per week.
* Currently uses tobacco or nicotine containing products, including but not limited to cigarettes, electronic cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum.
* Reported history of a significant traumatic injury, major surgery, or open biopsy within the 4 weeks prior to signing the informed consent form.
* Subject reported history of any use of long-term use of opioids agonists or antagonists; e.g., methadone, oxycodone, hydrocodone, naltrexone, buprenorphine.
* Subject reported history of any medications to treat opioid use disorder (MOUD); e.g., methadone, naltrexone, buprenorphine, kratom.
* Subject reports anticipated need for opioid analgesia in the next 12 months (e.g., planned surgery).
* Subject reports history or presence of allergic or adverse response (including rash or anaphylaxis) to naloxone, naltrexone, nalmefene, morphinan opioid agonists, benzyl alcohol or sesame oil.
* Positive urine drug screen (UDS) for barbiturates, benzodiazepines, cocaine, methamphetamine, or opioids.
* Positive alcohol breath test.
* Received an investigational drug within the last 30 days or 5 half-lives of the drug, whichever is longer, prior to administration of study medication.
* Has taken exclusionary prohibited medications within the last 30 days or 5 half-lives of the drug, whichever is longer.
* Subjects with a history of syncope, or have a history of symptomatic hypotension or symptomatic hypoglycemia.
* Subjects who test positive for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HbsAg), or Hepatitis C virus (HCV) antibody.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) | From predose through end of study visit, assessed up to study completion, an average of 15 months
  Number of Participants with TEAEs
Severity of TEAEs | From predose through end of study visit, assessed up to study completion, an average of 15 months
  Severity of TEAEs
Serious Adverse Events (SAEs) | From predose through end of study visit, assessed up to study completion, an average of 15 months
  Number of Participants with SAEs
Discontinuation Due to Adverse Events (AEs) | From predose through end of study visit, assessed up to study completion, an average of 15 months
  Number of Participants who discontinue the study due to AEs
Pharmacokinetics: AUC0-last | From predose through end of study visit, assessed up to study completion, an average of 15 months
  Area under the plasma concentration-time curve (AUC) from time 0 to last measurable plasma concentration
Pharmacokinetics: AUC0-infinity | From predose through end of study visit, assessed up to study completion, an average of 15 months
  Area under the plasma concentration-time curve from time 0 to infinity, calculated as AUC0-last + AUCt-inf
Pharmacokinetics: AUC0-inf %extrapolation | From predose through end of study visit, assessed up to study completion, an average of 15 months
  Percentage of AUC0-inf due to extrapolation from Tlast to infinity
Pharmacokinetics: Cmax | From predose through end of study visit, assessed up to study completion, an average of 15 months
  Maximum observed plasma concentration (Cmax)
Pharmacokinetics: Tmax | From predose through end of study visit, assessed up to study completion, an average of 15 months
  Time of Cmax
Pharmacokinetics: t1/2 | From predose through end of study visit, assessed up to study completion, an average of 15 months
  Terminal half-life (t1/2)
Pharmacokinetics: Kel (λz) | From predose through end of study visit, assessed up to study completion, an average of 15 months
  Apparent terminal rate-constant, calculated using linear regression on the terminal portion of the Log-concentration versus time curve
Pharmacokinetics: Vz/F | From predose through end of study visit, assessed up to study completion, an average of 15 months
  Apparent volume of distribution (Vz/F)
Pharmacokinetics: CL/F | From predose through end of study visit, assessed up to study completion, an average of 15 months
  Apparent clearance (CL/F)

CONTACTS AND LOCATIONS:
Overall Officials: N Shah, MD, Study Director — Nirsum Labs
Locations (1):
- Frontage Clinical Research Center, Secaucus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No